CLINICAL TRIAL: NCT01061307
Title: An Efficacy Trial of Fe, Zn and Vitamin A Fortified Rice in Children in Satun, Thailand
Brief Title: An Efficacy Trial of Iron, Zinc and Vitamin A Fortified Rice in Children in Satun, Thailand
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ETH2010/1
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2012-04

CONDITIONS: Vitamin A Deficiency; Iron Deficiency; Zinc Deficiency
Keywords: Fe deficiency, Zn deficiency, vitamin A deficiency
MeSH Terms: conditions — Vitamin A Deficiency; Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- fortified extruded rice (Experimental): fortified extruded rice (Fe, Zn and vitamin A) at the ratio 1:50 with normal rice
  Interventions: Dietary Supplement: fortified extruded rice

INTERVENTIONS:
Dietary Supplement: fortified extruded rice — fortified extruded rice (Fe, Zn and vitamin A) at the ratio 1:50 with normal rice

SUMMARY:
Iron, zinc and vitamin A deficiencies are particularly common among children and young women in the developing countries of South and Southeast Asia resulting in important adverse health effects. Simultaneous fortification of rice with iron, zinc and vitamin A could be a novel and sustainable approach to control these deficiencies.

Recently conducted extrusion trials have demonstrated that extruded rice grains containing iron, zinc and vitamin A show acceptable stability during production and storage and good sensory properties. The grains were produced using a twin-screw extruder equipped with a special cutter and a rice shaping die. The Fe, Zn and vitamin A content of the extruded product is 10 mg, 9 mg and 1050 μg per g of rice, respectively.

In this study the investigators plan to test the efficacy of the extruded triple fortified rice in Satun, Thailand, an area where rice is the staple food. Preliminary data from this area show that zinc and vitamin A intakes are low. Biochemical indicators have confirmed zinc deficiency and suboptimal vitamin A status in 1/3 of school aged children. The efficacy of the fortified rice will be evaluated in a 9 months, controlled, double-blind intervention trial in 7-12 y-old children. Children will be selected from primary schools in Satun Province based on low serum zinc values as the primary goal is to investigate Zn efficacy. As secondary outcome the effect on iron and vitamin A status will be investigated. The children will be randomized into two groups: a control group will receive a daily non-fortified rice lunch meal at school, while the second group will receive a daily rice meal containing the triple fortified rice. The rice meals will be given 5 days a week. At baseline, weight and height will be measured and determination of hemoglobin, serum ferritin, zinc protoporphyrin, serum zinc, serum retinol and C-reactive protein will be done. At mid-point and at 9 months, the baseline measurements will be repeated to judge the efficacy of the triple fortified rice.

ELIGIBILITY:
Inclusion Criteria:

* Preliminary screening: 650 children of 7-12 y-old children attending the primary school serving a low-income area in Muang district , Satun.(no exclusion criteria).
* Efficacy trial: 180-200 children, children with the Zn deficiency (serum zinc < 65, 66 and 70 µg/dL in children < 10y, male ≥ 10y and female ≥ 10y)

Exclusion Criteria:

* Children showing severe iron, zinc or vitamin A deficiency. These children will be excluded from the study and treated according to local policies.
* Significant chronic medical illness, including gastrointestinal, hematological, hepatic or renal disorders.
* Low school attendance (<80%).

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 203 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
serum Zn | September 2009-March 2010
Hemoglobin | September 2009-2010
serum retinol | September 2009-March 2010
serum ferritin | September 2009-March 2010
ZPP | September 2009- March 2010

SECONDARY OUTCOMES:
Anthropometry measures | September 2009-March 2010

CONTACTS AND LOCATIONS:
Locations (2):
- Swiss Federal Institute of Technology Zurich, Zurich, Switzerland
- Institute of Nutrition Mahidol University, Phuttamonthon, Changwat Nakhon Pathom, Thailand

REFERENCES:
- [Derived] Suri DJ, Tanumihardjo JP, Gannon BM, Pinkaew S, Kaliwile C, Chileshe J, Tanumihardjo SA. Serum retinol concentrations demonstrate high specificity after correcting for inflammation but questionable sensitivity compared with liver stores calculated from isotope dilution in determining vitamin A deficiency in Thai and Zambian children. Am J Clin Nutr. 2015 Nov;102(5):1259-65. doi: 10.3945/ajcn.115.113050. Epub 2015 Oct 7. PMID 26447158
- [Derived] Pinkaew S, Winichagoon P, Hurrell RF, Wegmuller R. Extruded rice grains fortified with zinc, iron, and vitamin A increase zinc status of Thai school children when incorporated into a school lunch program. J Nutr. 2013 Mar;143(3):362-8. doi: 10.3945/jn.112.166058. Epub 2013 Jan 9. PMID 23303870